CLINICAL TRIAL: NCT01558778
Title: Pilot Study of Mechanical Stimulation for Prevention of Hematopoietic Cell Transplant Associated Bone Density Loss
Brief Title: Mechanical Stimulation in Preventing Bone Density Loss in Patients Undergoing Donor Stem Cell Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: device not available
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 190510; NCI-2011-02354 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Neutrophilic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Disseminated Neuroblastoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Plasma Cell Neoplasm; Poor Prognosis Metastatic Gestational Trophoblastic Tumor; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Malignant Testicular Germ Cell Tumor; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Neuroblastoma; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage II Ovarian Epithelial Cancer; Stage II Ovarian Germ Cell Tumor; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Malignant Testicular Germ Cell Tumor; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Ovarian Epithelial Cancer; Stage III Ovarian Germ Cell Tumor; Stage III Small Lymphocytic Lymphoma; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Breast Cancer; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Neoplasms, Plasma Cell; Primary Myelofibrosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Testicular Neoplasms; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Neuroblastoma; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Breast Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (whole body vibration) (Experimental): Patients undergo mechanical stimulation over 20 minutes QD beginning on date of hospital admission and continuing through day 100 post-HCT, except for day 0 (date of transplant).
  Interventions: Procedure: management of therapy complications; Procedure: musculoskeletal complications management/prevention

INTERVENTIONS:
Procedure: management of therapy complications — Undergo mechanical stimulation
  Other Names: complications of therapy, management of
Procedure: musculoskeletal complications management/prevention — Undergo mechanical stimulation
  Other Names: complications management/prevention, musculoskeletal; management/prevention, musculoskeletal complications

SUMMARY:
This pilot clinical trial studies mechanical stimulation in preventing bone density loss in patients undergoing donor stem cell transplant. Mechanical stimulation may limit, prevent, or reverse bone loss, increase muscle and cardiac performance, and improve overall health

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of a mechanical stimulation regimen in hematopoietic cell transplant (HCT) patients.

SECONDARY OBJECTIVES:

I. To evaluate the data collection tools to prepare for a larger phase II trial.

OUTLINE:

Patients undergo mechanical stimulation over 20 minutes once daily (QD) beginning on date of hospital admission and continuing through day 100 post-HCT, except for day 0 (date of transplant).

ELIGIBILITY:
Inclusion Criteria:

* Meet eligibility criteria for first allogeneic HCT, and are scheduled to undergo allogeneic HCT
* Pre-transplant Karnofsky Performance Status (KPS) >= 70
* Patient or legal representative must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Any prior allogeneic HCT
* Pre-transplant weight >= 280 lbs
* Body mass index (BMI) < l8kg/m^2
* Human leukocyte antigen (HLA)-mismatched HCT
* Cord blood transplant
* Osteopenia or osteoporosis (T-score =< -1.0)
* Multiple myeloma diagnosis
* Any prior history of a central nervous system (CNS) hemorrhage
* Currently treated with a therapeutic dose of anti-coagulation for a recent pulmonary embolism or deep vein thrombosis
* Current or previous bisphosphonate use
* Prior history of non-traumatic fracture
* Any screws, pins, rods, or other metal objects in the body
* Total joint replacement
* History of kidney stones or gall stones
* Any artificial limbs
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Refinement of mechanical stimulation protocol | From hospital admission to 100 days post-HCT
  Best time of day for treatment, staff involvement, etc.
Adherence with treatment | From hospital admission to 100 days post-HCT
Effective data collection tools and data points | From hospital admission to 100 days post-HCT

CONTACTS AND LOCATIONS:
Overall Officials: Philip McCarthy, Principal Investigator — Roswell Park Cancer Institute